CLINICAL TRIAL: NCT06108375
Title: Differences in Acceptability of Music Therapy Sessions Played Live Compared to a Recording Thereof
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSIC
Record Dates: First submitted 2023-09-19; First posted 2023-10-31 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Terminal Illness; Terminal Cancer
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: monocentric study utilizing a prospective repeated measures design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live then recording (Other): During the first visit music will be played live, during the second visit a recording will play.
  Interventions: Other: music therapy; Other: recording
- Recording then live (Other): During the first visit a recording will play, during the second visit music will be played live.
  Interventions: Other: music therapy; Other: recording

INTERVENTIONS:
Other: music therapy — music played live by a music therapist
Other: recording — a recording of the same music played by the music therapist

SUMMARY:
The present study seeks to assess differences in feasibility and acceptability of music therapy played live and listening to a recording thereof at the palliative care ward of the University Hospital Zurich. As a secondary objective the investigators aim to extend the limited findings on the putative effect of music therapy in palliative care populations derived from objective measures of human autonomic response combined with subjective psychological outcomes to support evidence-based medicine. The investigators will implement a commercially available tracker, the wristband 287-2 by Corsano, to investigate multiple simultaneous biomarkers of autonomic response to music therapy and a recording thereof, such as heart rate, heart rate variability, electrodermal activity and distal body temperature.

To investigate subjective quality of life and psychological outcomes, the investigators will administer highly validated and widely used questionnaires, namely the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire 15 Palliative Care, the Edmonton Symptom Assessment System and the Hospital Anxiety and Depression Scale.

DETAILED DESCRIPTION:
The power of music to raise the spirits and to heal the soul should not be underestimated. There is growing recognition of the significance of music as a complementary treatment in palliative care, which is reflected in the growing body of scientific literature on the subject and in the popularly of music therapy among palliative care patients themselves.

Palliative care describes the holistic approach in the treatment of patients with advanced or incurable diseases, such as terminal cancer. In addition to conventional medical and nursing care, critical psychological, social and spiritual support is provided in palliative care. To this end, an interdisciplinary team of doctors, nursing staff, physiotherapists, occupational therapists, social workers, psycho-oncologists, chaplains and music therapists is involved.

Music therapy is defined as "the systematic use of music within a therapeutic relationship which aims at restoring, maintaining and furthering emotional, physical and mental health". The aim of music therapy in palliative care, in contrast, is to relieve symptoms of distress and improve quality of life among patients in the advanced stages of oncological disease. In Germany, national oncological guidelines currently recommend music therapy as a treatment option to alleviate anxiety and existential fear.

Music therapy encompasses both active and receptive techniques. Active techniques involve the patient in the production of music, such that they sing or play a musical instrument, possibly making planned gifts of songs to loved ones or for memorial services, whereas receptive techniques guide the patient in listening to music, both prerecorded as well as performed for them live. In cancer patients, the focus is placed primarily on music-assisted relaxation, generation of imagery, songs and improvisation. This heterogeneity of techniques studied in the literature on music therapy precludes an understanding of precisely what aspects of music therapy are most beneficial. Despite a diversity of approach, findings are promising, which in itself may be an indication as to whether the whole of music therapy is perhaps greater than the sum of its parts.

To practice music therapy according to the standards of evidence-based medicine, it is necessary to specify the intervention performed as well as the musical instrument(s) used. Moderators such as individual patient preferences and experience with music also may play an appreciable role; however, these are rarely systematically investigated.

Music therapy is conventionally administered by a trained music therapist and individual therapy sessions typically last 20 minutes. Training backgrounds of therapists vary, whereby in the United States a bachelor's degree in music therapy is the minimum requirement and board certification must follow in order for professional practice.

Few studies have investigated the efficacy of music therapy in palliative care patients. An emerging body of scientific literature in this clinical population suggests that music therapy may alleviate physical pain as well as psychological, social and emotional suffering. Spiritual needs may particularly benefit from music therapy.

Furthermore, a meta-analysis could show significant positive effects of music therapy on psychological wellbeing, physical symptoms and overall quality of life. Music therapy may favour various routine overarching themes in palliative care as well, such as pain management, relaxation, joy, hope, intensified spirituality and improved quality of life and may reduce anxiety and depression. Music therapy may outperform verbal exercises in inducing relaxation and reducing fatigue but not pain.

Despite the generally promising findings suggesting a benefit to psychological well-being assessed by subjective methods (e.g., visual analog scales, questionnaires, etc.) there is scant evidence derived from experiments utilizing objective outcome measures (e.g., autonomic response, etc.) with rigorous study design to support the efficacy of music therapy.

Findings derived from autonomic data suggest a benefit of music therapy characterized by increased parasympathetic tone accompanying improved subjective ratings of relaxation. Boosted high-frequency heart rate (HR) oscillations coincided with subjective relaxation score from visual analog scale after music therapy. In addition, blood volume pulse amplitude (BVP-A) was increased from baseline to post-therapy, indicating heightened vascular dilation due to greater parasympathetic activation, although just below the threshold of statistical significance (p = 0.07). In another analysis in the same sample, during music therapy higher levels of parasympathetically-mediated HR variability (HRV) were observed. Resting HR and blood pressure (BP) were reduced, whereas relaxation, comfort and happiness were increased. Increases in distal body temperature was observed in a sample of individuals undergoing chemotherapy. Anxiety related to chemotherapy was reduced by music therapy in this sample.

The present study seeks to assess differences in feasibility and acceptability of music therapy played live and listening to a recording thereof at the palliative care ward of the University Hospital Zurich. As a secondary objective the investigators aim to extend the limited findings on the putative effect of music therapy in palliative care populations derived from objective measures of human autonomic response combined with subjective psychological outcomes to support evidence-based medicine. The investigators will implement a commercially available tracker, the wristband 287-2 by Corsano, to investigate multiple simultaneous biomarkers of autonomic response to music therapy and a recording thereof, such as heart rate, heart rate variability, electrodermal activity and distal body temperature.

To investigate subjective quality of life and psychological outcomes, the investigators will administer highly validated and widely used questionnaires, namely the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire 15 Palliative Care, the Edmonton Symptom Assessment System and the Hospital Anxiety and Depression Scale.

The proposed risk category of this study is A. Justification for this risk categorization is reflected in the safe and relatively low burden of the study design, which requires the participants to undergo music therapy, complete questionnaires and wear a small wristwatch-like apparatus for a few minutes. Moreover, compared to conventional clinical measurement of human autonomic response, which typically involves skin disinfection and abrading followed by application of adhesive electrodes, the 287-2 wristband by Corsano is comparatively far less invasive and therefore represents diminished burden for the patient during their participation in the study. Music therapy and questionnaires (EORTC QLQ-C15-PAL, ESAS and HADS) are routine tasks for palliative care patients and represent no significant additional burden. In addition, the EORTC QLQ-C15-PAL questionnaire is the validated short-form version of the EORTC QLQ-C30-PAL, whose design objective is reduced patient burden. Furthermore, music therapy and these questionnaires are the standard of care in palliative care. The investigators submit that risk category A is appropriate given these methodological and ethical considerations.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Capacity to provide informed consent
* Patients with established diagnosis of a metastatic cancer/severe illness with limited life expectancy on a palliative care ward at the University Hospital Zurich

Exclusion Criteria:

• Inability to answer a questionnaire due to physical limitations as well as cognitive or linguistic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
intervention-specific acceptability questionnaire based on Theoretical Framework of Acceptability | immediately before and after the intervention
  assesses intervention acceptability, values 8 - 40, higher = better outcome

SECONDARY OUTCOMES:
Edmonton Symptom Assessment System | immediately before and after the intervention
  Assesses subjective symptom severity, values 0 - 120, higher = worse outcome
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire 15 Palliative Care | immediately before and after the intervention
  Assesses subjective quality of life, values 15 - 63, higher = worse outcome
Hospital Anxiety and Depression Scale | immediately before and after the intervention
  Assesses subjective anxiety and depression, values 0 - 42, higher = worse outcome
Qualitative open questions for patients | immediately before and after the intervention
  Assesses subjective experience of the intervention
Heart rate | immediately before and after the intervention
  Heart rate (bpm) is a basic marker of autonomic response and can reflect mortality and disease
Heart rate variability | immediately before and after the intervention
  Heart rate variability reflects neuro cardiac regulatory capacity and is a strong prognostic marker of mortality and disease
Electrodermal activity (μS; skin conductance response) | immediately before and after the intervention
  Electrodermal activity is a reliable biomarker of arousal
Temperature | immediately before and after the intervention
  Thermoregulation is tightly controlled and reacts to vigilance state

CONTACTS AND LOCATIONS:
Overall Officials: David Blum, Prof.Dr.med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No